CLINICAL TRIAL: NCT01343706
Title: A Randomized, Double-blind, Placebo-controlled (Within Dose Groups) Phase I Study to Assess Safety, Tolerability and Pharmacokinetics of Single Rising Doses 0.5 mg to 500 mg of BI 409306 Administered Orally in Healthy Male Volunteers
Brief Title: Safety Tolerability and Pharmacokinetic of BI 409306
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1289.1; 2010-023604-27 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-04-06; First posted 2011-04-28 (Estimated); Results first posted 2024-03-12 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Healthy
MeSH Terms: interventions — BI 409306

ARMS (12):
- BI 409306 0.5 mg PiB [EM] (Experimental): Extensive metaboliser [EM] subjects administered one single dose of 0.5 milligram (mg) BI 409306 powder in bottle (PiB) reconstituted for oral solution (0.5 mg /milliliter (mL)) in a volume of 80 mL of the solvent containing aqueous 0.5% tartaric acid solution orally with 240 mL water (160 mL containing the respective diluted volume of reconstituted solution and 80 mL drinking water) after an overnight fast of at least 10 hours.
  Interventions: Drug: BI 409306
- BI 409306 2 mg PiB [EM] (Experimental): EM subjects administered one single dose of 2 mg BI 409306 PiB reconstituted for oral solution (0.5 mg/mL) in a volume of 80 mL of the solvent containing aqueous 0.5% tartaric acid solution orally with 240 mL water (160 mL containing the respective diluted volume of reconstituted solution and 80 milliliter drinking water) after an overnight fast of at least 10 hours.
  Interventions: Drug: BI 409306
- BI 409306 5 mg PiB followed by BI 409306 5 mg Tablet [EM] (Experimental): EM subjects administered one single dose of 5 mg BI 409306 powder in bottle (PiB) reconstituted for oral solution (0.5 mg/ mL) in a volume of 80 mL of the solvent containing aqueous 0.5% tartaric acid solution orally with 240 mL water (160 mL containing the respective diluted volume of reconstituted solution and 80 mL drinking water) after an overnight fast of at least 10 hours in period 1; followed by a washout period of 5 days; followed by one single dose of 5 mg BI 409306 immediate release tablet administered orally with 240 mL water after an overnight fast of at least 10 hours in period 2.
  Interventions: Drug: BI 409306
- BI 409306 10 mg Tablet [EM] (Experimental): EM subjects administered 2 immediate release tablets of 5 mg BI 409306 as a single dose (total dosage: 10 mg) orally with 240 mL water after an overnight fast of at least 10 hours.
  Interventions: Drug: BI 409306
- BI 409306 25 mg Tablet [EM] (Experimental): EM subjects administered 5 immediate release tablets of 5 mg BI 409306 as a single dose (total dosage: 25 mg) orally with 240 mL water after an overnight fast of at least 10 hours.
  Interventions: Drug: BI 409306
- BI 409306 50 mg Tablet followed by BI 409306 50mg PiB [EM] (Experimental): EM subjects administered one single dose of 50 mg BI 409306 immediate release tablet orally with 240 mL water in period 1; followed by a washout period of 5 days; followed by one single dose of 50 mg BI 409306 powder in bottle (PiB) reconstituted for oral solution (0.5 mg/mL) in a volume of 80 mL of the solvent containing aqueous 0.5% tartaric acid solution administered orally with 240 mL water (160 mL containing the respective diluted volume of reconstituted solution and 80 mL drinking water) after an overnight fast of at least 10 hours in period 2.
  Interventions: Drug: BI 409306
- BI 409306 100 mg Tablet [EM] (Experimental): EM subjects administered 2 immediate release tablets of 50 mg BI 409306 as single dose (total dosage: 100 mg) orally with 240 mL water after an overnight fast of at least 10 hours.
  Interventions: Drug: BI 409306
- BI 409306 200 mg Tablet [EM] (Experimental): EM subjects administered 1 immediate release tablet of 150 mg and 1 immediate release tablet of 50 mg of BI 409306 together as single dose (total dosage: 200 mg) orally with 240 mL water after an overnight fast of at least 10 hours.
  Interventions: Drug: BI 409306
- BI 409306 350 mg Tablet [EM] (Experimental): EM subjects administered 2 immediate release tablet of 150 mg and 1 immediate release tablet of 50 mg of BI 409306 together as single dose (total dosage: 350 mg) orally with 240 mL water after an overnight fast of at least 10 hours.
  Interventions: Drug: BI 409306
- BI 409306 10 mg Tablet followed by BI 409306 100mg Tablet [PM] (Experimental): Poor metaboliser [PM] subjects administered 2 immediate release tablets of 5 mg BI 409306 as single dose (total dosage: 10 mg) orally with 240 mL water after an overnight fast of at least 10 hours in period 1; followed by washout period of 5 days; followed by 2 immediate release tablets of 50 mg BI 409306 administered as single dose (total dosage: 100 mg) orally with 240 mL water after an overnight fast of at least 10 hours in period 2.
  Interventions: Drug: BI 409306
- Placebo matching to BI 409306 PiB (Placebo Comparator): Subjects administered one single dose of placebo matching to BI 409306 powder in bottle (PiB) after an overnight fast of at least 10 hours.
  Interventions: Drug: Placebo
- Placebo matching to BI 409306 film-coated tablet (Placebo Comparator): Subjects administered one single dose of placebo matching to the BI 409306 film-coated tablet (5 milligrams (mg), 50 mg, and 150 mg) orally with 240 mL water after an overnight fast of at least 10 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Solution for oral administration
  Arms: Placebo matching to BI 409306 PiB
Drug: Placebo — Immediate release solid oral dosage (film-coated tablet)
  Arms: Placebo matching to BI 409306 film-coated tablet
Drug: BI 409306 — Immediate release solid oral dosage (film-coated tablet)
  Arms: BI 409306 10 mg Tablet [EM]; BI 409306 10 mg Tablet followed by BI 409306 100mg Tablet [PM]; BI 409306 100 mg Tablet [EM]; BI 409306 200 mg Tablet [EM]; BI 409306 25 mg Tablet [EM]; BI 409306 350 mg Tablet [EM]; BI 409306 5 mg PiB followed by BI 409306 5 mg Tablet [EM]; BI 409306 50 mg Tablet followed by BI 409306 50mg PiB [EM]
Drug: BI 409306 — solution for oral administration
  Arms: BI 409306 0.5 mg PiB [EM]; BI 409306 2 mg PiB [EM]; BI 409306 5 mg PiB followed by BI 409306 5 mg Tablet [EM]; BI 409306 50 mg Tablet followed by BI 409306 50mg PiB [EM]

SUMMARY:
The primary objective of the current study is to investigate the safety and tolerability of BI 409306 in healthy male genotyped volunteers following oral administration of single rising doses.

The secondary objectives are: (1) to explore dose proportionality of BI 409306 as immediate release solid oral dosage, (2) to explore the relative bioavailability of BI 409306 when administered as immediate release solid oral dosage compared to oral drinking solution and (3) to compare the safety and pharmacokinetic profiles between two different groups of genotyped subjects.

ELIGIBILITY:
Inclusion criteria:

1. Healthy males according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), clinical laboratory tests
2. Age > 21 and Age < 50 years
3. Body Mass Index (BMI) > 18.5 and BMI < 29.9 kg/m2

Exclusion criteria:

1. Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
2. Any evidence of a clinically relevant concomitant disease
3. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
4. Surgery of the gastrointestinal tract (except appendectomy)
5. Diseases of the central nervous system (including but not limited to any kind of seizures, stroke or psychiatric disorders) within the past 6 month
6. History of relevant orthostatic hypotension, fainting spells or blackouts.
7. Chronic or relevant acute infections
8. History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
9. Use of drugs which might reasonably influence the results of the trial or that prolong the QT/QTc interval based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
10. Any laboratory value outside the reference range that is of clinical relevance
11. A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms);
12. A history of additional risk factors for Torsades de points (TdP) (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2011-04-01 (Actual); Primary Completion 2011-08-01 (Actual); Study Completion 2011-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1289.1.1 Boehringer Ingelheim Investigational Site, Ingelheim, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this Phase 1, single centre, placebo-controlled trial (within dose groups), total of 80 healthy subjects were entered and 79 (71 CYP2C19 Extensive metaboliser /8 Poor CYP2C19 metaboliser) subjects were treated in 10 sequential dose groups.
Pre-assignment Details: All subjects were screened for eligibility to participate in the trial. Subjects attended specialist sites which would then ensure that all subjects met all inclusion/exclusion criteria. Subjects were not to be randomised to trial treatment if any one of the specific entry criteria were not met.
Groups:
- Placebo Matching to BI 409306 [EM and PM]: Extensive metaboliser [EM] subjects administered one single dose of placebo matching to BI 409306 powder in bottle (PiB) reconstituted for oral solution or one single dose of placebo matching to BI 409306 tablet orally with 240 mL water after an overnight fast of at least 10 hours.
  Poor metaboliser [PM] subjects administered one single dose of placebo matching to BI 409306 powder in bottle (PiB) reconstituted for oral solution or one single dose of placebo matching to BI 409306 tablet orally with 240 mL water after an overnight fast of at least 10 hours in period 1; followed by a washout period of 5 days; followed by one single dose of placebo to BI 409306 tablet administered orally with 240 mL water after an overnight fast of at least 10 hours in period 2.
- Placebo to BI 409306 50 mg Tablet Followed by BI 409306 50 mg PiB [EM]: EM subject administered one single dose of placebo matching to the 50 mg BI 409306 film-coated tablet orally with 240 mL water in period 1; followed by a washout period of 5 days; followed by 50 mg BI 409306 powder in bottle (PiB) reconstituted for oral solution administered orally with 240 mL water in period 2, both after an overnight fast of at least 10 hours.
Period: Overall Study
Arm/Group | Placebo Matching to BI 409306 [EM and PM] | BI 409306 0.5 mg PiB [EM] | BI 409306 2 mg PiB [EM] | BI 409306 5 mg PiB Followed by BI 409306 5 mg Tablet [EM] | BI 409306 10 mg Tablet [EM] | BI 409306 25 mg Tablet [EM] | BI 409306 50 mg Tablet Followed by BI 409306 50mg PiB [EM] | Placebo to BI 409306 50 mg Tablet Followed by BI 409306 50 mg PiB [EM] | BI 409306 100 mg Tablet [EM] | BI 409306 200 mg Tablet [EM] | BI 409306 350 mg Tablet [EM] | BI 409306 10 mg Tablet Followed by BI 409306 100mg Tablet [PM]
Started (Entered subjects) | 18 | 6 | 6 | 6 | 6 | 6 | 6 | 2 | 6 | 6 | 6 | 6
Not Treated (Subject withdrew before the first drug administration) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Completed (Completed planned observation time) | 18 | 6 | 6 | 6 | 6 | 6 | 6 | 2 | 5 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The treated set includes all subjects who were dispensed study medication and were documented to have taken at least one dose of investigational treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Matching to BI 409306 [EM and PM] | BI 409306 0.5 mg PiB [EM] | BI 409306 2 mg PiB [EM] | BI 409306 5 mg PiB Followed by BI 409306 5 mg Tablet [EM] | BI 409306 10 mg Tablet [EM] | BI 409306 25 mg Tablet [EM] | BI 409306 50 mg Tablet Followed by BI 409306 50mg PiB [EM] | Placebo to BI 409306 50 mg Tablet Followed by BI 409306 50 mg PiB [EM] | BI 409306 100 mg Tablet [EM] | BI 409306 200 mg Tablet [EM] | BI 409306 350 mg Tablet [EM] | BI 409306 10 mg Tablet Followed by BI 409306 100mg Tablet [PM] | Total
Number analyzed (Participants) | 18 | 6 | 6 | 6 | 6 | 6 | 6 | 2 | 5 | 6 | 6 | 6 | 79
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at the time of signing informed consent form is presented. Population: TS
  Years | 38.2 (5.6) | 36.5 (9.2) | 37.5 (6.5) | 35.7 (8.2) | 30.5 (5.9) | 32.2 (6.5) | 40.3 (6.1) | 37.5 (3.5) | 31.4 (7.3) | 38.5 (6.7) | 39.2 (8.8) | 39.5 (7.5) | 36.7 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Number of subjects is categorized as Male or Female. Population: TS
  Participants
    Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Male | 18 | 6 | 6 | 6 | 6 | 6 | 6 | 2 | 5 | 6 | 6 | 6 | 79
Race (NIH/OMB) [Count of Participants; unit: Participants] — Number of subjects is categorized for race data. Ethnicity data were not collected. Population: TS
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    White | 18 | 6 | 6 | 6 | 6 | 6 | 6 | 2 | 5 | 6 | 6 | 6 | 79
    More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Drug-related Adverse Events
Description: Percentage of subjects with investigator defined drug-related Adverse Events (AEs)
Time Frame: From first drug administration until 30 days after last drug administration; up to 31 days.
Population: Treated set (TS):This set includes all subjects who were dispensed study medication and were documented to have taken at least one dose of investigational treatment.
Measure: Number; unit: Percentage of subjects
Groups:
- Placebo Matching to BI (Period 1): Extensive metaboliser [EM] and poor metaboliser [PM] subjects randomized to placebo treatment (in period 1 only, if having 2 periods).
- Placebo Matching to BI (Period 2): Extensive metaboliser [EM] and poor metaboliser [PM] subjects administered placebo in period 2 (after a wash out period of 5 days).
- BI 409306 5 mg PiB [EM]: EM subjects administered one single dose of 5 mg BI 409306 powder in bottle (PiB) reconstituted for oral solution (0.5 mg/ mL) in a volume of 80 mL of the solvent containing aqueous 0.5% tartaric acid solution orally with 240 mL water (160 mL containing the respective diluted volume of reconstituted solution and 80 mL drinking water) after an overnight fast of at least 10 hours in period 1.
- BI 409306 5 mg Tablet [EM]: EM subjects administered one single dose of 5 mg BI 409306 immediate release tablet administered orally with 240 mL water after an overnight fast of at least 10 hours in period 2 (after a washout period of 5 days).
- BI 409306 10 mg Tablet [EM]: Subjects administered 2 single doses of 10 mg BI 409306 immediate release tablets orally with 240 mL water after an overnight fast of at least 10 hours in extensive metabolizer [EM] group.
- BI 409306 25 mg Tablet [EM]: Subjects administered a single dose of 25 mg BI 409306 immediate release tablets orally with 240 mL water after an overnight fast of at least 10 hours in extensive metabolizer [EM] group.
- BI 409306 50 mg Tablet [EM]: EM subjects administered one single dose of 50 mg BI 409306 immediate release tablet orally with 240 mL water in period 1.
- BI 409306 50 mg PiB [EM]: Subjects administered one single dose 50 ml BI 409306 powder in bottle (PiB) reconstituted for oral solution (0.5 ml/mL) in a volume of 80 mL of the solvent containing aqueous 0.5% tartaric acid solution orally with 240 mL water (160 mL containing the respective diluted volume of reconstituted solution and 80 mL drinking water) after washout period of 5 days both after an overnight fast of at least 10 hours in extensive metabolizer [EM] group.
- BI 409306 100 mg Tablet [EM]: Subjects administered 2 single doses of 100 mg BI 409306 immediate release tablets orally with 240 mL water after an overnight fast of at least 10 hours in extensive metabolizer [EM] group.
- BI 409306 200 mg Tablet [EM]: Subjects administered a single dose of 200 mg BI 409306 immediate release tablets orally with 240 mL water after an overnight fast of at least 10 hours in extensive metabolizer [EM] group.
- BI 409306 350 mg Tablet [EM]: Subjects administered a single dose of 350 mg BI 409306 immediate release tablets orally with 240 mL water after an overnight fast of at least 10 hours in extensive metabolizer [EM] group.
- BI 409306 10 mg Tablet [PM]: Poor metaboliser [PM] subjects administered 2 immediate release tablets of 5 mg BI 409306 as single dose (total dosage: 10 mg) orally with 240 mL water after an overnight fast of at least 10 hours in period 1.
- BI 409306 100 mg Tablet [PM]: PM subjects administered 2 immediate release tablets of 50 mg BI 409306 as single dose (total dosage: 100 mg) orally with 240 mL water after an overnight fast of at least 10 hours in period 2 (after a washout period of 5 days).
Arm/Group | Placebo Matching to BI (Period 1) | Placebo Matching to BI (Period 2) | BI 409306 0.5 mg PiB [EM] | BI 409306 2 mg PiB [EM] | BI 409306 5 mg PiB [EM] | BI 409306 5 mg Tablet [EM] | BI 409306 10 mg Tablet [EM] | BI 409306 25 mg Tablet [EM] | BI 409306 50 mg Tablet [EM] | BI 409306 50 mg PiB [EM] | BI 409306 100 mg Tablet [EM] | BI 409306 200 mg Tablet [EM] | BI 409306 350 mg Tablet [EM] | BI 409306 10 mg Tablet [PM] | BI 409306 100 mg Tablet [PM]
Number analyzed (Participants) | 20 | 4 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 5 | 6 | 6 | 6 | 6
Percentage of subjects | 0.0 | 0.0 | 0.0 | 33.3 | 0.0 | 16.7 | 0.0 | 0.0 | 0.0 | 0.0 | 40.0 | 66.7 | 66.7 | 33.3 | 50.0

2. Primary Outcome: Percentage of Subjects With Clinical Relevant Abnormalities for Physical Examination, Vital Signs, Clinical Laboratory Tests, Oral Body Temperature and ECG
Description: Percentage of subjects with Clinical Relevant abnormalities for Physical examination, Vital Signs blood pressure (BP), pulse rate (PR) respiratory rate (RR), orthostatic test), Clinical laboratory tests (haematology, clinical chemistry and urinalysis), Oral body temperature and ECG were reported.
Time Frame: Day 4
Population: as for outcome 1
Measure: Number; unit: Percentage of subjects
Groups:
- BI 409306 5 mg Tablet EM: Subjects administered a single dose of 5 mg BI 409306 immediate release tablets orally with 240 mL water after an overnight fast of at least 10 hours and after washout period of 5 days in extensive metabolizer [EM] group.
- BI 409306 50 mg Tablet [EM]: Subjects administered one single dose of 50 mg BI 409306 immediate release tablets orally with 240 mL water after washout period of 5 days both after an overnight fast of at least 10 hours in extensive metabolizer [EM] group.
- BI 409306 10 mg Tablet [PM]: Subjects administered 2 single doses of 10 mg film-coated tablet of BI 409306 orally with 240 mL water after an overnight fast of at least 10 hours in poor metabolizer [PM] group.
- BI 409306 100 mg Tablet [PM]: Subjects administered 2 single doses of 100 mg film-coated tablet of BI 409306 orally with 240 mL water after an overnight fast of at least 10 hours in poor metabolizer [PM] group.
Arm/Group | Placebo Matching to BI (Period 1) | Placebo Matching to BI (Period 2) | BI 409306 0.5 mg PiB [EM] | BI 409306 2 mg PiB [EM] | BI 409306 5 mg PiB [EM] | BI 409306 5 mg Tablet EM | BI 409306 10 mg Tablet [EM] | BI 409306 25 mg Tablet [EM] | BI 409306 50 mg Tablet [EM] | BI 409306 50 mg PiB [EM] | BI 409306 100 mg Tablet [EM] | BI 409306 200 mg Tablet [EM] | BI 409306 350 mg Tablet [EM] | BI 409306 10 mg Tablet [PM] | BI 409306 100 mg Tablet [PM]
Number analyzed (Participants) | 20 | 4 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 5 | 6 | 6 | 6 | 6
Percentage of subjects | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Percentage of Subjects Per Category for Assessment of Tolerability by Investigator
Description: The investigator assessed global clinical assessment and tolerability of BI 409306 were reported in possible categories were 'good', 'satisfactory', 'not satisfactory', and 'bad'.
Time Frame: Day 4
Population: as for outcome 1
Measure: Number; unit: Percentage of subjects
Groups:
- BI 409306 25 mg Tablet [EM]: Subjects were administered a single dose of 25 mg BI 409306 immediate release tablets orally with 240 mL water after an overnight fast of at least 10 hours.
- BI 409306 350 mg Tablet [EM]: Subjects administered a single dose of 350 mg BI 409306 immediate release tablets orally with 240 mL water after an overnight fast of at least 10 hours.
Arm/Group | Placebo Matching to BI 409306 [EM and PM] | BI 409306 0.5 mg PiB [EM] | BI 409306 2 mg PiB [EM] | BI 409306 5 mg PiB Followed by BI 409306 5 mg Tablet [EM] | BI 409306 10 mg Tablet [EM] | BI 409306 25 mg Tablet [EM] | BI 409306 50 mg Tablet Followed by BI 409306 50mg PiB [EM] | Placebo to BI 409306 50 mg Tablet Followed by BI 409306 50 mg PiB [EM] | BI 409306 100 mg Tablet [EM] | BI 409306 200 mg Tablet [EM] | BI 409306 350 mg Tablet [EM] | BI 409306 10 mg Tablet Followed by BI 409306 100mg Tablet [PM]
Number analyzed (Participants) | 18 | 6 | 6 | 6 | 6 | 6 | 6 | 2 | 5 | 6 | 6 | 6
Percentage of subjects
  Good | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 2 | 5 | 6 | 4 | 4
  Satisfactory | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
  Not satisfactory | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Bad | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not assessable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Change From Baseline in Bond & Lader (B&L) Visual Analogue Scales (VAS)
Description: The B&L VAS scores were calculated from 16 item with each has a score range from 0 to 10 [cm]. The score of each of the 3 categories of effects ("alertness", "calmness", and "contentment") is a weighted average of the scores from the 16 items. The VAS score for alertness/calmness/contentment ranges from 0 to 10 (more alertness/calmness/contentment). The B&L VAS data was analysed descriptively (change from baseline at 24 hour). The VAS assessment 2 h before drug administration was considered as baseline.
Time Frame: At 24 hours
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo Matching to BI (Period 1) | Placebo Matching to BI (Period 2) | BI 409306 0.5 mg PiB [EM] | BI 409306 2 mg PiB [EM] | BI 409306 5 mg PiB [EM] | BI 409306 5 mg Tablet [EM] | BI 409306 10 mg Tablet [EM] | BI 409306 25 mg Tablet [EM] | BI 409306 50 mg Tablet [EM] | BI 409306 50 mg PiB [EM] | BI 409306 100 mg Tablet [EM] | BI 409306 200 mg Tablet [EM] | BI 409306 350 mg Tablet [EM] | BI 409306 10 mg Tablet [PM] | BI 409306 100 mg Tablet [PM]
Number analyzed (Participants) | 20 | 4 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 5 | 6 | 6 | 6 | 6
Score on a scale
  Alertness | -0.33 (1.26) | -0.04 (0.70) | -0.84 (1.11) | -1.18 (0.35) | -0.13 (0.70) | 0.09 (0.56) | -0.33 (0.73) | -0.07 (0.97) | -0.92 (1.25) | -0.56 (0.54) | -0.26 (0.95) | -0.80 (0.55) | -0.21 (0.39) | -1.02 (1.24) | -1.88 (1.58)
  Contentment | -0.30 (1.09) | 0.06 (0.45) | -0.74 (1.02) | -0.68 (0.23) | -0.53 (0.68) | -0.12 (0.71) | 0.04 (0.46) | 0.00 (0.76) | -0.49 (0.84) | -0.35 (0.75) | -0.19 (0.73) | -0.59 (0.59) | -0.22 (0.50) | -0.64 (1.23) | -0.97 (0.71)
  Calmness | -0.35 (1.34) | 0.02 (0.21) | -0.48 (1.20) | -0.91 (0.99) | -0.45 (0.89) | -0.14 (1.59) | 0.25 (1.04) | -0.39 (0.55) | -0.75 (1.35) | -0.47 (1.71) | 0.05 (1.31) | -0.55 (1.55) | -0.17 (0.34) | -0.47 (1.06) | -0.38 (0.59)

5. Secondary Outcome: Area Under the Concentration-time Curve of the BI 409306 in Plasma From Time 0 to Time of Last Quantifiable Data Point (AUC0-24)
Description: AUC0-24, Area under the concentration-time curve of the BI 409306 in plasma over the time interval from 0 to the time of the last quantifiable data point is presented as geometric mean (gMean) and geometric coefficient of variation (gCV%). Pharmacokinetic samples were also collected at 48:00 and 72:00 hours after the drug administration for dose groups 10 mg onwards.
Time Frame: Pharmacokinetic samples were collected at 2:00 (hour: minute) before 0.167, 0.333, 0.5, 0.75, 1:00, 1.50, 2:00, 2.50, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 14:00, and 24:00 hours after the drug administration.
Population: Per protocol set for evaluation of PK (PPS-PK): This set included all evaluable subjects of the treated set who had no important protocol violations relevant to the evaluation of PK, who had no pre-dose value greater than 5% of Cmax and who did not vomit or had diarrhoea at or before two times median tmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol*hour/Litre [nmol*h/L]
Arm/Group | BI 409306 0.5 mg PiB [EM] | BI 409306 2 mg PiB [EM] | BI 409306 5 mg PiB [EM] | BI 409306 5 mg Tablet [EM] | BI 409306 10 mg Tablet [EM] | BI 409306 25 mg Tablet [EM] | BI 409306 50 mg Tablet [EM] | BI 409306 50 mg PiB [EM] | BI 409306 100 mg Tablet [EM] | BI 409306 200 mg Tablet [EM] | BI 409306 350 mg Tablet [EM] | BI 409306 10 mg Tablet [PM] | BI 409306 100 mg Tablet [PM]
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 5 | 6 | 6 | 6 | 6
nanomol*hour/Litre [nmol*h/L] | 3.96 (50.3) | 20.90 (41.30) | 76.70 (27.00) | 75.60 (32.29) | 96.00 (69.90) | 351.00 (49.30) | 539.00 (82.00) | 648.00 (42.90) | 1460.00 (68.50) | 3920.00 (44.40) | 7980.00 (17.10) | 476.00 (35.40) | 6060.00 (21.40)

6. Secondary Outcome: Area Under the Concentration-time Curve of the BI 409306 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: AUC0-∞, Area under the concentration-time curve of the BI 409306 in plasma over the time interval from 0 extrapolated to infinity. Pharmacokinetic samples were also collected at 48:00 and 72:00 hours after the drug administration for dose groups 10 mg onwards.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol*hour/Litre [nmol*h/L]
Arm/Group | BI 409306 0.5 mg PiB [EM] | BI 409306 2 mg PiB [EM] | BI 409306 5 mg PiB [EM] | BI 409306 5 mg Tablet [EM] | BI 409306 10 mg Tablet [EM] | BI 409306 25 mg Tablet [EM] | BI 409306 50 mg Tablet [EM] | BI 409306 50 mg PiB [EM] | BI 409306 100 mg Tablet [EM] | BI 409306 200 mg Tablet [EM] | BI 409306 350 mg Tablet [EM] | BI 409306 10 mg Tablet [PM] | BI 409306 100 mg Tablet [PM]
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 5 | 6 | 6 | 6 | 6
nanomol*hour/Litre [nmol*h/L] | 3.95 (50.40) | 20.90 (41.30) | 76.70 (27.00) | 75.60 (32.20) | 95.90 (69.80) | 351.00 (49.40) | 539.00 (82.00) | 648.00 (42.90) | 1460.00 (68.50) | 3920.00 (44.40) | 7980.00 (17.10) | 476.00 (35.50) | 6060.00 (21.40)

7. Secondary Outcome: Maximum Measured Concentration of the BI 409306 in Plasma (Cmax)
Description: Cmax, Maximum measured concentration of the BI 409306 in plasma. Pharmacokinetic samples were also collected at 48:00 and 72:00 hours after the drug administration for dose groups 10 mg onwards.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol/Litre (nmol/L)
Arm/Group | BI 409306 0.5 mg PiB [EM] | BI 409306 2 mg PiB [EM] | BI 409306 5 mg PiB [EM] | BI 409306 5 mg Tablet [EM] | BI 409306 10 mg Tablet [EM] | BI 409306 25 mg Tablet [EM] | BI 409306 50 mg Tablet [EM] | BI 409306 50 mg PiB [EM] | BI 409306 100 mg Tablet [EM] | BI 409306 200 mg Tablet [EM] | BI 409306 350 mg Tablet [EM] | BI 409306 10 mg Tablet [PM] | BI 409306 100 mg Tablet [PM]
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 5 | 6 | 6 | 6 | 6
nanomol/Litre (nmol/L) | 3.54 (34.50) | 18.80 (50.80) | 56.40 (36.40) | 55.90 (40.90) | 99.80 (79.10) | 300.00 (85.00) | 479.00 (67.00) | 613.00 (40.70) | 1370.00 (87.30) | 2950.00 (89.50) | 5540.00 (29.50) | 223.00 (38.10) | 3120.00 (31.40)

8. Secondary Outcome: Amount of BI 409306 Eliminated in Urine From the Time Point t1 to Time Point t2 (Ae0-4)
Description: Ae0-4, Amount of BI 409306 eliminated in urine from the time point t1(0) to time point t2(4). Urine samples were obtained 24:00 to 48:00 and 48:00 to 72:00 hours after oral administration were obtained only from dose group 10 mg onwards.
Time Frame: Urine samples were obtained pre-dose and sampling intervals 0:00 to 4:00, 4:00 to 8:00, 8:00 to 12:00 and 12:00 to 24:00 hours after oral administration.
Population: Per protocol set for evaluation of PK (PPS-PK): This set included all evaluable subjects of the treated set who had no important protocol violations relevant to the evaluation of PK, who had no pre-dose value greater than 5% of Cmax and who did not vomit or had diarrhoea at or before two times median tmax. Only participants with non-missing outcomes were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol [nmol]
Arm/Group | BI 409306 0.5 mg PiB [EM] | BI 409306 2 mg PiB [EM] | BI 409306 5 mg PiB [EM] | BI 409306 5 mg Tablet [EM] | BI 409306 10 mg Tablet [EM] | BI 409306 25 mg Tablet [EM] | BI 409306 50 mg Tablet [EM] | BI 409306 50 mg PiB [EM] | BI 409306 100 mg Tablet [EM] | BI 409306 200 mg Tablet [EM] | BI 409306 350 mg Tablet [EM] | BI 409306 10 mg Tablet [PM] | BI 409306 100 mg Tablet [PM]
Number analyzed (Participants) | 0 | 6 | 6 | 6 | 5 | 0 | 6 | 8 | 4 | 5 | 6 | 6 | 6
nanomol [nmol] |  | 31.00 (46.50) | 93.60 (26.00) | 98.10 (24.20) | 148.00 (60.20) |  | 840.00 (56.90) | 953.00 (48.10) | 1920.00 (53.00) | 4340.00 (48.80) | 8830.00 (24.00) | 418.00 (14.30) | 5700.00 (23.30)

ADVERSE EVENTS:
Time Frame: From first drug administration until 30 days after last drug administration; up to 31 days.
Description: The safety analysis was based on treated set (TS). TS includes all subjects who were dispensed study medication and were documented to have taken at least one dose of investigational treatment.
Groups:
- BI 409306 50mg PiB [EM]: EM subjects administered one single dose of 50 mg BI 409306 powder in bottle (PiB) reconstituted for oral solution (0.5 mg/mL) in a volume of 80 mL of the solvent containing aqueous 0.5% tartaric acid solution orally with 240 mL water (160 mL containing the respective diluted volume of reconstituted solution and 80 mL drinking water) after an overnight fast of at least 10 hours in period 2 (after a washout period of 5 days).
Arm/Group | Placebo Matching to BI (Period 1) | Placebo Matching to BI (Period 2) | BI 409306 0.5 mg PiB [EM] | BI 409306 2 mg PiB [EM] | BI 409306 5 mg PiB [EM] | BI 409306 5 mg Tablet [EM] | BI 409306 10 mg Tablet [EM] | BI 409306 25 mg Tablet [EM] | BI 409306 50 mg Tablet [EM] | BI 409306 50mg PiB [EM] | BI 409306 100 mg Tablet [EM] | BI 409306 200 mg Tablet [EM] | BI 409306 350 mg Tablet [EM] | BI 409306 10 mg Tablet [PM] | BI 409306 100 mg Tablet [PM]
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/4 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/8 | 0/5 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/4 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/8 | 0/5 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 2/20 | 1/4 | 0/6 | 2/6 | 0/6 | 1/6 | 0/6 | 0/6 | 2/6 | 0/8 | 2/5 | 4/6 | 4/6 | 3/6 | 3/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo Matching to BI (Period 1) (N=20) | Placebo Matching to BI (Period 2) (N=4) | BI 409306 0.5 mg PiB [EM] (N=6) | BI 409306 2 mg PiB [EM] (N=6) | BI 409306 5 mg PiB [EM] (N=6) | BI 409306 5 mg Tablet [EM] (N=6) | BI 409306 10 mg Tablet [EM] (N=6) | BI 409306 25 mg Tablet [EM] (N=6) | BI 409306 50 mg Tablet [EM] (N=6) | BI 409306 50mg PiB [EM] (N=8) | BI 409306 100 mg Tablet [EM] (N=5) | BI 409306 200 mg Tablet [EM] (N=6) | BI 409306 350 mg Tablet [EM] (N=6) | BI 409306 10 mg Tablet [PM] (N=6) | BI 409306 100 mg Tablet [PM] (N=6)
Extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0/5 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Chromatopsia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Photopsia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes